CLINICAL TRIAL: NCT02488109
Title: Multi-center Randomized Controlled Trial of Refeeding in Anorexia Nervosa
Brief Title: Study of Refeeding to Optimize iNpatient Gains
Acronym: StRONG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Stanford University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P0504491; 1R01HD082166-01A1 (NIH); NCT02621229 (obsolete NCT alias)
Record Dates: First submitted 2015-06-23; First posted 2015-07-02 (Estimated); Results first posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Anorexia Nervosa
Keywords: anorexia nervosa; eating disorders; refeeding; adolescent medicine; nutritional rehabilitation
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Higher Calorie Refeeding Protocol (Active Comparator): Participants in this arm will receive a higher calorie meal-based refeeding treatment plan in hospital.
  Interventions: Other: Higher Calorie Refeeding
- Lower Calorie Refeeding Protocol (Active Comparator): Participants in this arm will receive a lower calorie meal-based refeeding treatment plan in hospital.
  Interventions: Other: Lower Calorie Refeeding

INTERVENTIONS:
Other: Higher Calorie Refeeding
  Arms: Higher Calorie Refeeding Protocol
Other: Lower Calorie Refeeding
  Arms: Lower Calorie Refeeding Protocol

SUMMARY:
The purpose of this study is to compare the efficacy, safety, and cost-effectiveness of lower calorie refeeding versus higher calorie refeeding in hospitalized adolescents with anorexia nervosa.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of AN
* atypical AN
* no hospital admissions for the previous six months
* meet hospitalization criteria: daytime heart rate (HR) < 50 bpm or night time HR < 45 bpm, blood pressure (BP) <90/45 mmHg, temperature < 35.6° C, or symptomatic orthostasis defined by increase in HR > 35 bpm or decrease in systolic BP > 20 mmHg or decrease in diastolic BP > 10 mmHg from lying to standing

Exclusion Criteria:

* diagnosis of bulimia nervosa [DSM-5]
* currently in remission (as defined by weight and EDE-Q score)
* admission for food refusal without malnutrition
* current pregnancy
* chronic disease (e.g. immune/endocrine disorders, pulmonary, cardiac, or renal disease)
* current suicidality or psychosis
* < 60% mBMI

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea K Garber, PhD, RD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Stanford University Lucille Packard Children's Hospital, Palo Alto, California
  - University of California, San Francisco Benioff Children's Hospital, San Francisco, California

REFERENCES:
- [Derived] Vendlinski SS, Gorrell S, Downey AE, Mehta AS, Le Grange D, Machen VI, Accurso EC, Buckelew SM, Kapphahn CJ, Moscicki BA, Golden NH, Garber AK. Self-Reported Physical Activity Energy Expenditure in Patients With Anorexia Nervosa: A Cross-Sectional Analysis at Hospital Admission From the Study of Refeeding to Optimize iNpatient Gains. Int J Eat Disord. 2026 Jan;59(1):122-133. doi: 10.1002/eat.24569. Epub 2025 Oct 6. PMID 41047835
- [Derived] Golden NH, Cheng J, Kapphahn CJ, Buckelew SM, Machen VI, Kreiter A, Accurso EC, Adams SH, Le Grange D, Moscicki AB, Sy AF, Wilson L, Garber AK. Higher-Calorie Refeeding in Anorexia Nervosa: 1-Year Outcomes From a Randomized Controlled Trial. Pediatrics. 2021 Apr;147(4):e2020037135. doi: 10.1542/peds.2020-037135. Epub 2021 Mar 22. PMID 33753542
- [Derived] Garber AK, Cheng J, Accurso EC, Adams SH, Buckelew SM, Kapphahn CJ, Kreiter A, Le Grange D, Machen VI, Moscicki AB, Sy A, Wilson L, Golden NH. Short-term Outcomes of the Study of Refeeding to Optimize Inpatient Gains for Patients With Anorexia Nervosa: A Multicenter Randomized Clinical Trial. JAMA Pediatr. 2021 Jan 1;175(1):19-27. doi: 10.1001/jamapediatrics.2020.3359. PMID 33074282
- [Derived] Garber AK, Cheng J, Accurso EC, Adams SH, Buckelew SM, Kapphahn CJ, Kreiter A, Le Grange D, Machen VI, Moscicki AB, Saffran K, Sy AF, Wilson L, Golden NH. Weight Loss and Illness Severity in Adolescents With Atypical Anorexia Nervosa. Pediatrics. 2019 Dec;144(6):e20192339. doi: 10.1542/peds.2019-2339. Epub 2019 Nov 6. PMID 31694978

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from February 8, 2016, to March 7, 2019 at 2 clinical sites, large tertiary care children's hospitals with eating disorder inpatient programs attended by interdisciplinary adolescent medicine care teams at the University of California San Francisco and Stanford University. Written informed consent was obtained from young adults and parents of minors, who provided written assent.
Pre-assignment Details: Although 120 participants were randomized,116 started on the study. Of the 4 individuals who were randomized but did not receive treatment, 3 were found ineligible and 1 did not complete the consent, leaving 56 individuals in the LCR arm. Of those 56 individuals, an additional 5 individuals withdrew prior to receiving treatment, ultimately resulting in 51 participants in the LCR arm.
Groups:
- Higher Calorie Refeeding (HCR) Protocol: Meal-based refeeding in hospital: starting 2000 kcal/d and increasing 200 kcal/d to goal
- Lower Calorie Refeeding (LCR) Protocol: Meal-based refeeding in hospital: starting 1400 kcal/d and increasing 200 kcal every other day to goal
Period: Treatment in Hospital
Arm/Group | Higher Calorie Refeeding (HCR) Protocol | Lower Calorie Refeeding (LCR) Protocol
Started | 60 | 56
Received Treatment | 60 | 51
Included in mITT Analysis | 60 | 51
Completed | 60 | 51
Not Completed | 0 | 5
Not completed — Withdrawal by Subject | 0 | 5
Period: 12-month Follow-Up
Arm/Group | Higher Calorie Refeeding (HCR) Protocol | Lower Calorie Refeeding (LCR) Protocol
Started (Discharge from hospital) | 60 | 51
Included in mITT Analysis | 60 | 51
Completed (Retained in trial through 12 months) | 56 | 44
Not Completed | 4 | 7
Not completed — Lost to Follow-up | 4 | 7

BASELINE CHARACTERISTICS:
Population: Modified Intention to Treat Analysis (mITT) includes all participants who received treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Higher Calorie Refeeding (HCR) Protocol | Lower Calorie Refeeding (LCR) Protocol | Total
Number analyzed (Participants) | 60 | 56 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.6 (2.5) | 16.2 (2.4) | 16.4 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 52 | 105
  Male | 7 | 4 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Non-Hispanic White | 36 | 33 | 69
  Race/ethnicity: Asian | 7 | 7 | 14
  Race/ethnicity: Hispanic or Latino | 15 | 9 | 24
  Race/ethnicity: Other or >1 race/ethnicity reported | 2 | 7 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60 | 56 | 116
Admission percentage of median body mass index (%mBMI) [Mean (Standard Deviation); unit: % of mBMI] | 83.3 (11.1) | 86.6 (12.2) | 84.6 (11.9)
Lowest 24-hr heart rate, beats/min [Mean (Standard Deviation); unit: beats per minute] | 41.5 (6.9) | 40.7 (5.9) | 41.3 (6.1)
Lowest Systolic Blood Pressure (mm Hg) [Mean (Standard Deviation); unit: mm Hg] | 94.2 (8.0) | 93.3 (8.3) | 93.7 (8.1)
Global Eating Disorder Examination Questionnaire score (mean, SD) [Mean (Standard Deviation); unit: Score on a scale] — Scores range from 1-6, with higher scores indicating greater severity. For reference, the EDE-Q global score in community studies is 3.38.
  Score on a scale | 3.32 (1.68) | 3.45 (1.71) | 3.34 (1.70)
Atypical anorexia nervosa (No., %) [Count of Participants; unit: Participants] | 21 | 27 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Remission at Different Time Points of Assessment
Description: Clinical remission was defined as the combination of percentage mBMI and EDE-Q score at 1, 3, 6, and 12 months. This is a dichotomous variable 1/0. If participants achieve both weight recovery (defined as =>95% of median BMI for sex and age), AND psychological recovery (defined as within 1SD of community norms for EDE-Q) then they are assigned a "1" for achieving clinical remission. If both parameters not met then "0" for not remitted.
Time Frame: up to 12 months
Population: Clinical remission defined as the combination of %mBMI and EDE-Q score. Instead of assuming missing data at random in the generalized linear mixed-effects regression model, clinical remission was modeled as a nominal multinomial outcome (yes, no, or missing), with time (1, 3, 6, or 12 months after discharge), treatment group, and time*treatment group interaction as fixed effects. Longitudinal analysis included only participants with both %mBMI and EDE-Q scores.
Measure: Count of Participants; unit: Participants
Arm/Group | Higher Calorie Refeeding (HCR) Protocol | Lower Calorie Refeeding (LCR) Protocol
Number analyzed (Participants) | 44 | 34
Participants
  1 month: number analyzed (Participants) | 40 | 32
  1 month | 12 | 8
  3 months: number analyzed (Participants) | 39 | 34
  3 months | 10 | 13
  6 months: number analyzed (Participants) | 39 | 26
  6 months | 16 | 10
  12 months: number analyzed (Participants) | 44 | 27
  12 months | 18 | 13
Statistical Analysis 1: Comparison: Higher Calorie Refeeding (HCR) Protocol vs Lower Calorie Refeeding (LCR) Protocol; The study was powered to detect a difference in 12-months clinical remission rates between groups. N = 60 per arm with 85% retention would provide 80% power on a 2-sided 0.05-level test to detect a 20% difference between groups in 12-months clinical remission rates. A generalized linear mixed-effects regression model was used to compare study arms with respect to achievement and maintenance of clinical remission; Test type: Other; p = 0.42, Regression, Linear — Changes in rates of clinical remission by group over time in the mITT model; Clinical remission was modeled as a nominal multinomial outcome (yes, no, or missing)

2. Secondary Outcome: Time to Achieve Medical Stability in Hospital
Description: Medical stability was adjudicated by a 6-point clinical index: (1) 24-hour heart rate of 45 beats/min or more, (2) systolic blood pressure of 90 mm Hg or more, (3) temperature of 35.6 °C or more, (4) orthostatic increase in heart rate of 35 beats/min or less, (5) orthostatic decrease in systolic blood pressure of 20 mm Hg or less, and (6) 75% or more of mBMI for age and sex. Criteria were assessed daily; for vital signs with multiple daily measures, the most deviant value was recorded (eg, lowest heart rate). Each criterion was scored as "1" if met, "0" if unmet, and missing (not scored) if not measured. Medical stability was considered restored when all measured criteria were stable for 24 hours, allowing a maximum of 2 missing values. Additional efficacy outcomes were time to restore heart rate to 45 beats/min or more (among those with bradycardia at baseline) and weight gain (change in percentage mBMI).
Time Frame: Inpatient hospitalization from day of admission to day of discharge, average of 10 days
Population: Modified intention to treat analysis (mITT) included all participants who received at least one day of treatment
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Higher Calorie Refeeding (HCR): Meal-based refeeding in hospital: starting 2000 kcal/d and increasing 200 kcal/d to goal
- Lower Calorie Refeeding (LCR): Meal-based refeeding in hospital: starting 1400 kcal/d and increasing 200 kcal every other day to goal
Arm/Group | Higher Calorie Refeeding (HCR) | Lower Calorie Refeeding (LCR)
Number analyzed (Participants) | 60 | 51
Days | 7.0 (7.0) | 10.0 (8.0)
Statistical Analysis 1: Comparison: Higher Calorie Refeeding (HCR) vs Lower Calorie Refeeding (LCR); This trial was powered at 0.80 to detect a 12% to 20% difference in restored medical stability at 0.05 type I error and correlation between time points from 0.1 to 1; Test type: Superiority; p = 0.01, Survival analysis with log rank test — Survival analysis of time to medical stability by log-rank test, which does not assume proportional hazards. Those who did not reach medical stability before hospital discharge were censored; analyses accounted for the site effect by stratification; Compared time to achieve medical stability by arm; participants who did not meet stability criteria by hospital discharge were right-censored; Hazard Ratio (HR) = 1.67, 95% CI 2-sided [1.10 to 2.53]

3. Other Pre Specified Outcome: Cost-effectiveness Per Adolescent Recovered
Description: defined as total cost (direct and indirect costs)
Time Frame: up to 12 months
Population: The analysis was a modified intent-to-treat (mITT) approach including all randomized participants who received treatment for at least one day. A total of 9 participants were excluded: 3 were found to be ineligible after randomization and 6 withdrew prior to receiving treatment.
Measure: Median (Standard Deviation); unit: USD
Arm/Group | Higher Calorie Refeeding (HCR) Protocol | Lower Calorie Refeeding (LCR) Protocol
Number analyzed (Participants) | 60 | 51
USD | 38,112 (26,043) | 57,168 (30,486)
Statistical Analysis 1: Comparison: Higher Calorie Refeeding (HCR) Protocol vs Lower Calorie Refeeding (LCR) Protocol; Cost outcomes of group differences and 95% confidence intervals were estimated; Test type: Superiority; p = 0.002, Wilcoxon (Mann-Whitney); Median Difference (Net) = 19,056, 95% CI 2-sided [9,293 to 28,819]

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events on an ongoing basis during the treatment period, which was during hospitalization from day of admission to day of discharge (an average of 10 days). After the treatment effect window was completed on discharge from the hospital, adverse events were not considered to be related to study treatment.
Groups:
- Lower Calorie Refeeding (LCR): Meal-based refeeding in hospital: starting 1400 kcal/d and increasing 200 kcal every other day to goal. Of the 56 participants originally randomized to this treatment, 5 never received treatment and were therefore excluded from mITT analyses.
Arm/Group | Higher Calorie Refeeding (HCR) | Lower Calorie Refeeding (LCR)
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/51
Serious Adverse Events (participants affected / at risk) | 14/60 | 10/51
Other Adverse Events (participants affected / at risk) | 14/60 | 21/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Higher Calorie Refeeding (HCR) (N=60) | Lower Calorie Refeeding (LCR) (N=51)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) — <2.5 mg/dL
Orthostatic increase in heart rate (Metabolism and nutrition disorders) | 4 (20) | 4 (16) — An increase in heart rate from lying (for 5 min) to standing (for 2 min) was categorized as severe in this patient population if it reached a threshold of a change of >75 bpm
Psychiatric SAE, e.g. suicide attempt (Psychiatric disorders) | 3 (4) | 3 (3) — All of these psychiatric events occurred during the follow-up period, after patients were no longer in our care
Severe Bradycardia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — <30 bpm
Severe Hypotension (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — <80/40
Other unrelated SAEs during follow-up period (Metabolism and nutrition disorders) | 6 (6) | 0 (0) — e.g. elevated liver enzymes, sialolithiasis, gallstone pancreatitis, renal calculi, tonic clonic seizure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Higher Calorie Refeeding (HCR) (N=60) | Lower Calorie Refeeding (LCR) (N=51)
Hypokalemia (mild) (Metabolism and nutrition disorders) | 3 (4) | 5 (5) — 3.1 - 3.4 mmol/L
Hypomagnesemia (mild) (Metabolism and nutrition disorders) | 7 (10) | 14 (16) — 1.3 - 1.7 mg/dL
Hypophosphatemia (moderate) (Metabolism and nutrition disorders) | 4 (4) | 2 (2) — Moderate: 2.5 - 2.9 mg/dL

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/09/NCT02488109/Prot_SAP_000.pdf